CLINICAL TRIAL: NCT03356405
Title: Evaluating Treatment as Prevention Among People Who Inject Drugs in Dundee for HCV
Acronym: ERAPID HCV
Status: Active, not recruiting | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, John Dillon, Professor John Dillon, University of Dundee
Other Study IDs: 2016GA08
Record Dates: First submitted 2017-11-17; First posted 2017-11-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hepatitis C Viral
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to conduct an evaluation of hepatitis C treatments in NHS Tayside in order to empirically test the "treatment as prevention" models. This will be done by analysing the records of patients who have been tested and treated for hepatitis C using NHS Tayside databases. There will be no interventions carried out as part of this study.

DETAILED DESCRIPTION:
Hepatitis C is a blood-borne virus (HCV) that can seriously damage the liver and is spread mainly through blood-to-blood contact with an infected person. The "serious and significant public health risk" posed by HCV was recognised during a member's debate in the Scottish Parliament in 2004. By December 2006, Health Protection Scotland estimated that 50,000 persons in Scotland had been infected with the Hepatitis C virus and that 38,000 were chronic carriers. Currently, the greatest risk of acquiring the virus in the UK is through injecting drug use. In Scotland, it is estimated that over 85% of individuals who have Hepatitis C were infected in this way.

The outcome of HCV infection varies considerably between individuals. Some (up to 25%) are able to clear the infection spontaneously, whilst the remaining 75% become chronically infected. Within the subpopulation of chronically infected patients, some will develop serious liver disease, including cirrhosis and hepatocellular carcinoma, within a few years, whilst in others liver disease will not progress even over a period of more than forty years. Hepatitis C is often referred to as the 'silent epidemic.' Many who are infected are unaware of it, and often show no symptoms over a long period of time. While there is presently no vaccination for Hepatitis C, the recent introduction of protease inhibitor-based directly acting anti-viral treatments (DAA) has begun a new era in treatment of this disease. These new oral treatments are extremely safe, have shorter treatment regimens than previous drugs, and are effective, producing a cure in over 90% of cases providing compliance is adequate.

The advent of more effective DAA therapies raises the possibility of using therapy as prevention, turning the epidemic off at source, by targeting active infected drug users who are the main source of new infections.

The modelling work of the investigators shows that HCV treatment is a critical component to HCV prevention among people who inject drugs and is likely to be cost-effective compared to delaying treatment or treating non-PWID with mild or moderate disease. For example, the investigators show in a number of settings with chronic HCV in PWID below 60% that treating 10-20 per 1000 drug users per year can reduce HCV prevalence by 50-90% over 10-15 years; that for every one PWID treated in the 20% chronic HCV setting 2 new HCV infections are averted. The scale of the benefit is inversely and exponentially related to prevalence of HCV in the population, the lower the prevalence the sooner and bigger the impact.

Current conventional treatment pathways focus on populations drawn from those known to drug problem services and former drug users. Treating people who are the most stable and with a low risk of relapse back into chaotic injecting will reduce future morbidity in the individual patients but may not achieve additional benefit in terms of averting future infections. The recent work of the investigators within Tayside has shown that they are able to test less stable, actively injecting drug users for Hepatitis C and then successfully treat them using both the conventional care pathway and non-conventional care pathways, such as needle exchange clinics (e.g. Eradicate study, completed February 2017; Advance study, aiming to start in October 2017), community pharmacies (SuperDOTC study, ongoing) and prisons. If the models are correct, this intensive treatment programme will effectively eradicate Hepatitis C from Tayside over the next few years. However, the models are not yet empirically tested and they make some assumptions that if violated may lead to over or under-estimation of the intervention effect. For example, the models assume that (a) heterogeneity in injecting risk and uptake of HCV testing and treatment will even out as PWID move and transition between high and low risk periods; and (b) that HCV transmission risk for susceptible PWID is similar for those that have achieved SVR or are untreated.

The intensive treatment approach in Tayside provides an ideal opportunity to empirically test the "treatment as prevention" models. The current study will not involve direct recruitment or treatment of patients. Instead, it will evaluate the portfolio of care pathways currently being used to treat HCV in Tayside and test the hypothetical modelling to determine whether treatment of HCV will work as prevention of future spread of the virus.

ELIGIBILITY:
Inclusion Criteria:

* All individuals in NHS Tayside eligible for HCV testing and treatment according to Scottish Intercollegiate Guidelines Network guidelines.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals in NHS Tayside eligible for HCV testing and treatment according to Scottish Intercollegiate Guidelines Network guidelines.
Sampling Method: Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of HCV positive tests recorded in NHS Tayside. | 6 years
  The number of reactive DBST conducted in NHS Tayside.

SECONDARY OUTCOMES:
The number of patients engaged in treatment and SVR12 during the treatment phase | 6 years
  The numbers of patients who are treated for HCV and the number who achieve an SVR12.
The cost of treatment | 6 years
  The cost of treating HCV infection in PWID will be measured.
Re-infection with HCV following treatment | 6 years
  Annual routine offer of HCV testing

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Tayside, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03356405/Prot_SAP_000.pdf